CLINICAL TRIAL: NCT04494074
Title: Intérêt du Traitement de la fièvre Par Refroidissement Externe Pour la Survie Des Patients ventilés en Choc Septique
Brief Title: Fever Control Using External Cooling in Mechanically Ventilated Patients With Septic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEPSISCOOL II
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Septic Shock
Keywords: External cooling,; Fever; ARDS
MeSH Terms: conditions — Shock, Septic; Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fever Control by external cooling (Experimental): External cooling during 48 hours to obtain normothermia
  Interventions: Other: External Cooling
- Fever respected, no cooling (No Intervention): Fever respect without any antipyretic therapy

INTERVENTIONS:
Other: External Cooling — External Cooling
  Arms: Fever Control by external cooling

SUMMARY:
The best strategy for managing fever in patients with septic shock remains unknown. In a pilot study, the investigators showed that fever control at normothermia allowed a better control of shock and evolution of organ failures. In this second trial the investigators will conduct a multicentre, open-label, randomized controlled, superiority trial in which two strategies will be compared:

1. Respect of fever
2. Fever control at normothermia using external cooling The primary end point will be d-60 mortality.

DETAILED DESCRIPTION:
Sepsis is a common syndrome responsible for multiple organ failure. Septic shock, defined as sepsis with hyperlactatemia and cardiovascular failure requiring vasopressor infusion despite adequate fluid resuscitation has an extremely high mortality rate. Fever is a frequent disease process during sepsis. Fever increases oxygen consumption and can worsen imbalance between oxygen supply and oxygen requirements. Fever increases inflammation but reduces viral and bacterial growth. The beneficial effects of active fever control on inflammation have been mainly shown in a context of lung injury. Pneumonia represents the first cause of septic shock in developed countries.

In a pilot study (SEPSISCOOL I), we showed that fever treatment using external cooling significantly increased the resolution of shock, improved organ functions and decreased d-14 mortality. Although reduced, hospital mortality was not significantly different. This study was underpowered to allow conclusion on mortality. A more pronounced beneficial effect was observed among the most severely ill patients with elevated serum lactate level.

Fever treatment is commonly applied in septic patients but its impact on survival remains undetermined.

The main objective of the study is to compare two strategies of fever management in febrile (body temperature > 38.3°C) septic shock patients requiring invasive mechanical ventilation and sedation. These patients will be randomly allocated in two arms:

1. Fever respect
2. Fever control by external cooling to obtain normothermia during 48 hours

A covariate-adaptive randomization will be used to ensure the comparability of the two groups at each stage of the study. We will use an adaptive multistage population-enrichment design with a pre-specified subgroup of patients with ARDS identified at randomization.

An independent Safety and Data Monitoring Committee will review data on serious adverse events. The decision of study stop for potential harmful effect of one strategy will be let at the entire responsibility of the committee.

One interim analysis will be performed by independent observers after enrolment of half of the population. The assumption that fever treatment is more effective in patients with ARDS will be confirmed or not. According to pre-defined rules based on the conditional power calculated in the two subgroups, the trial will be stopped for futility, continued as planned or continued by enrolling only patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Documented or suspected infection either communautary or hospital acquired
* Septic shock defined by the need for vasopressor and lactate>2 mmol/l despite adequate fluid resuscitation (sepsis-3 definition)
* Patients under invasive mechanical ventilation
* Body core temperature>38.3°C
* Intravenous sedation or opioids
* Ongoing antimicrobial treatment and/or intervention for infection source control
* Attending physician confirms clinical equipoise without substantial risk if the patient participates in the trial
* Informed consent of next of kin/other designated person before inclusion or procedure for inclusion in emergency situation

Exclusion Criteria:

* Cardiac arrest within previous 7 days
* Acute brain injury within previous 7 days
* Extensive burns or epidermal necrolysis
* <18 years old
* Body core temperature >41°C
* Under legal guardianship
* No affiliation with the French health-care system
* Pregnancy
* Participation in another interventional study with mortality as the primary endpoint
* An investigator's decision not to resuscitate
* Patient already recruited in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Day 60 from randomization
  All causes mortality

SECONDARY OUTCOMES:
Evolution of SOFA Score | Up to Day 7
  Sequential Organ Failure Assessment (SOFA) score will be calculated at d1, d2, d3 and d7 and compared between the 2 arms.
  Higer the score higher the severity of organ dysfunctions. Min 0 Max 24
Number of ventilator free days | Day 28
  Number of free days will be assessed as proposed by YEHYA et al. Patients who died before d28 will be considered as having 0 free day
Number of renal replacement therapy free days | Day 28
  Number of free days will be assessed as proposed by YEHYA et al.
Number of vasopressor free days | Day 28
  Number of free days will be assessed as proposed by YEHYA et al. Shock resolution will be defined by vasopressor stop during at least 24h in the absence of care withdrawing
Mortality | Day 28
  All causes mortality
Number of patients with shivering | Day 2
  Shivering will be monitored according to a specific scale
Number of patients with seizure | Day 3
  Seizure will be clinically documented or reveal by EEG
Number of patients with hypothermia | Day 3
  Number of patients with body temperature lower than 36°C
Number of patients with at least 1 episode of cardiac arrhythmia | Day 3
  Patient with new episode of supraventricular or ventricular arrhythmia
Secondary acquired nosocomial infections | Day 28
  Only the first episode will be taken into account
Number of patients with ARDS development among patients free of ARDS at inclusion | Up to Day 3
  Secondary acquired ARDS according to Berlin definition
Acute kidney injury in patients free of RRT at inclusion | Up to Day7
  Maximal stage of AKI according to the KDIGO definition

CONTACTS AND LOCATIONS:
Locations (33):
- France (33):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - Hôpital Nord Franche Comté, Belfort
  - CH Cholet, Cholet
  - Centre hospitalier intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - CHD Dijon, Dijon
  - CHU Grenoble, Grenoble
  - GH Est Francilien, Jossigny
  - CHD Vendée, La Roche-sur-Yon
  - CHU Kremlin Bicetre, Le Kremlin-Bicêtre
  - CHU Le Mans, Le Mans
  - CH Lens, Lens
  - CH Libourne, Libourne
  - Hôpital Saint Joseph Saint Luc, Lyon
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Timone, Marseille
  - CHR Metz Hôpital de Mercy, Metz
  - GRH Mulhouse, Mulhouse
  - CHU Hotel Dieu, Nantes
  - CHU Archet 1, Nice
  - Hôpital Pasteur, Nice
  - Hopital Lariboisière - Réanimation Médicale, Paris
  - Hôpital Lariboisière -Réanimation chirurgicale, Paris
  - CHU La Milétrie Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Charles Nicolle, Rouen
  - CHU Réunion Sud, Saint-Denis
  - Hôpital FOCH, Suresnes
  - CH BIGORRE SITE GESPE Tarbes, Tarbes
  - CHBA Vannes-Auray, Vannes
  - Centre Hospitalier Mignot, Versailles

IPD SHARING:
Plan to Share IPD: Yes
Strictly anonymized data will be available upon justified request from the coordinating investigator and the study sponsor
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After publication upon justified request from the coordinating investigator and the study sponsor

REFERENCES:
- [Derived] Guenegou-Arnoux A, Murris J, Bechet S, Jung C, Auchabie J, Dupeyrat J, Anguel N, Asfar P, Badie J, Carpentier D, Chousterman B, Bourenne J, Delbove A, Devaquet J, Deye N, Dumas G, Dureau AF, Lascarrou JB, Legriel S, Guitton C, Janniere-Nartey C, Quenot JP, Lacherade JC, Maizel J, Mekontso Dessap A, Mourvillier B, Petua P, Plantefeve G, Richard JC, Robert A, Saccheri C, Vong LVP, Katsahian S, Schortgen F; REVA Network. Protocol for fever control using external cooling in mechanically ventilated patients with septic shock: SEPSISCOOL II randomised controlled trial. BMJ Open. 2024 Jan 29;14(1):e069430. doi: 10.1136/bmjopen-2022-069430. PMID 38286691